CLINICAL TRIAL: NCT04777331
Title: A Phase IIB, Randomized, Double-Blind, Placebo-Controlled, Multicenter Study to Evaluate the Efficacy and Safety of Intravenous Prasinezumab in Participants With Early Parkinson's Disease
Brief Title: A Study to Evaluate the Efficacy and Safety of Intravenous Prasinezumab in Participants With Early Parkinson's Disease
Acronym: PADOVA
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Prothena Biosciences Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BN42358; 2020-004997-23 (EudraCT Number); 2023-507132-21-00 (EU CTIS Number)
Record Dates: First submitted 2021-02-26; First posted 2021-03-02 (Actual); Results first posted 2025-12-02 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Parkinsons Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Prasinezumab (Experimental): Participants will receive an IV infusion of prasinezumab every 4 weeks (Q4W).
  Participants will enter into the optional Open Label Extension (OLE) once the double-blind treatment period has completed.
  Interventions: Drug: Prasinezumab
- Placebo (Placebo Comparator): Participants will receive placebo as an IV infusion Q4W.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Prasinezumab — Prasinezumab will be administered as an IV infusion to participants Q4W.
  Arms: Prasinezumab
Drug: Placebo — Prasinezumab placebo will be administered to participants.
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled study that will evaluate the efficacy and safety of intravenous (IV) prasinezumab versus placebo in participants with Early Parkinson's Disease (PD) who are on stable symptomatic PD medication.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic PD based on MDS criteria with bradykinesia plus one of the other cardinal signs of PD (resting tremor, rigidity), without any other known or suspected cause of parkinsonism
* On symptomatic PD medication, with stable doses for at least 3 months prior to baseline
* A diagnosis of PD for at least 3 months to maximum 3 years at screening
* MDS-UPDRS Part IV score of 0 at screening and prior to randomization
* Hoehn and Yahr (H&Y) Stage I or II in OFF medication state at screening and prior to randomization
* Dopamine transporter imaging with single photon emission computed tomography (DaT-SPECT) imaging consistent with dopamine transporter deficit, as assessed by the central reader
* No anticipated changes in PD medication from baseline throughout the study duration based on clinical status during screening
* Willingness and ability to use a smartphone application to measure PD-related symptoms for the duration of the study
* Willingness and ability to wear a smartwatch to measure PD-related motor signs

Exclusion Criteria:

* Medical history indicating a Parkinsonian syndrome other than idiopathic PD
* Diagnosis of PD dementia
* Diagnosis of a significant neurologic disease other than PD
* Within the last year, unstable or clinically significant cardiovascular disease
* Uncontrolled hypertension
* Drug and/or alcohol abuse within 12 months prior to screening, in the investigator's judgment (Nicotine is allowed, Marijuana use is not allowed)
* Clinically significant abnormalities in laboratory test results at the screening visit, including hepatic and renal panels, complete blood count, chemistry panel and urinalysis
* Allergy to any of the components of prasinezumab, a known hypersensitivity, or a previous IRR following administration of any other monoclonal antibody
* Any contraindications to obtaining a brain magnetic resonance imaging (MRI)
* Any contraindications to DaT-SPECT imaging

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 586 (Actual)
Dates: Start 2021-05-05 (Actual); Primary Completion 2024-09-11 (Actual); Study Completion 2026-12-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (110):
- United States (31):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Barrow Neurological Institute, Phoenix, Arizona
  - Neurology Center of North Orange County, Fullerton, California
  - UC San Diego, La Jolla, California
  - Keck School of Medicine of USC, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - CenExel Rocky Mountain Clinical Research, LLC, Englewood, Colorado
  - Institute for Neurodegenerative Disorders, New Haven, Connecticut
  - JEM Research LLC, Atlantis, Florida
  - Parkinson's Disease and Movement Disorders Center of Boca Raton, Boca Raton, Florida
  - Renstar Medical Research, Ocala, Florida
  - University of South Florida, Tampa, Florida
  - Charter Research - Winter Park/Orlando, Winter Park, Florida
  - Northwestern University Feinberg School Of Medicine, Chicago, Illinois
  - Southern Illinois University, School of Medicine, Springfield, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - Quest Research Institute, Farmington Hills, Michigan
  - Henry Ford Hospital, West Bloomfield, Michigan
  - Dent Neurological Institute, Amherst, New York
  - Cleveland Clinic, Cleveland, Ohio
  - The Movement Disorder Clinic of Oklahoma, Tulsa, Oklahoma
  - University Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Texas Neurology PA, Dallas, Texas
  - Baylor College of Medicine Medical Center, Houston, Texas
  - Central Texas Neurology Consultants, Round Rock, Texas
  - University of Vermont Medical Center, Burlington, Vermont
  - Sentara Neurology Specialists, Norfolk, Virginia
  - EvergreenHealth Investigational Drug Services, Kirkland, Washington
  - Inland Northwest Research, Spokane, Washington
- Austria (3):
  - Medizinische Universität Graz, Graz
  - Uniklinik fuer Neurologie, Medizinische Universitaet Innsbruck, Innsbruck
  - Klinik Ottakring, Vienna
- Canada (4):
  - Toronto Memory Program, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario
  - Clinique Neuro Outaouais, Gatineau, Quebec
  - Montreal Neurological Institute and Hospital, Montreal, Quebec
- France (15):
  - Groupe Hospitalier Pellegrin, Bordeaux
  - Groupement Hospitalier Est - Hôpital Neurologique, Bron
  - Hopital Gabriel Montpied, Clermont-Ferrand
  - Hôpital Henri Mondor, Créteil
  - Hôpital Michallon - Centre d'Investigation Clinique, Grenoble
  - CHU de Limoges - Hôpital Dupuytren, Limoges
  - hopital de la Timone, Marseille
  - CHU Gui de Chauliac, Montpellier
  - CHU de Nice Hopital Pasteur, Nice
  - Hopital Pitie-Salpetriere APHP, Paris
  - CHU Poitiers, Poitiers
  - CHU Rouen Charles Nicolle, Rouen
  - CHU de Nantes - Hopital Laennec, Saint-Herblain
  - CHU Strasbourg Hpital Hautepierre, Strasbourg
  - CIC - Hôpital Purpan, Toulouse
- Italy (15):
  - Università degli studi della Campania Luigi Vanvitelli, Napoli, Campania
  - Az. Osp. OO.RR. S. Giovanni di Dio e Ruggi D' Aragona, Salerno, Campania
  - Ospedale Bellaria, Bologna, Emilia-Romagna
  - IRCCS San Raffaele;Clinical Trial Center, Rome, Lazio
  - Policlinico Universitario Agostino Gemelli, Rome, Lazio
  - Irccs A.O.U.San Martino Ist, Genoa, Liguria
  - Azienda Ospedaliera Spedali Civili, Brescia, Lombardy
  - IRCCS Ospedale San Raffaele, Milan, Lombardy
  - IRCCS Istituto Neurologico Carlo Besta, Milan, Lombardy
  - IRCCS Neuromed, Pozzilli (IS), Molise
  - A.O.U. Policlinico "G.Rodolico - San Marco", Catania, Sicily
  - A.O. Universitaria Pisana, Pisa, Tuscany
  - AO di Perugia - Ospedale S. Maria della Misericordia, Perugia, Umbria
  - Azienda Ospedaliera S. Maria, Terni, Umbria
  - Azienda Ospedaliera di Padova, Padua, Veneto
- Centre Hospitalier de Luxembourg, Luxembourg, Luxembourg
- Poland (9):
  - NeuroKlinika Gabinet Lekarski Prof. Andrzej Bogucki, ?ód?
  - NZOZ Vitamed, Bydgoszcz
  - Szpital Sw. Wojciecha, Gda?sk
  - Krakowska Akademia Neurologii Sp z o.o. Centrum Neurologii K, Krakow
  - Indywidualna Praktyka Lekarska Prof. Dr Hab. N. Med. Konrad Rejdak., Lublin
  - Nmedis sp. z o.o., Rzeszów
  - Samodzielny Publiczny Szpital Kliniczny im. prof. Orlowskiego, Warsaw
  - Centrum Medyczne NeuroProtect, Warsaw
  - Mazowiecki Szpital Bródnowski w Warszawie Sp. z o.o., Warsaw
- Spain (25):
  - Hospital General Universitario de Elche, Elche, Alicante
  - Hospital General De Catalunya, Sant Cugat del Vallès, Barcelona
  - Policlínica Guipuzkoa, Donosti-San Sebastián, Guipuzcoa
  - Complejo Hospitalario Universitario A Coruña (CHUAC), A Coruña, LA Coruna
  - Hospital Universitario Fundación Alcorcón, Alcorcón, Madrid
  - HM Universitario Puerta del Sur CINAC (C.Integ.Neuroc);, Móstoles, Madrid
  - Hospital Quiron de Madrid, Pozuelo de Alarcón, Madrid
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Hospital Virgen del Puerto, Plasencia, Palencia
  - Hospital de Cruces, Barakaldo, Vizcaya
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Clinic Servicio de Neurologia, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario de Burgos. Servicio de Neurología, Burgos
  - Hospital Ruber Juan Bravo, Madrid
  - Hospital Universitario de la Princesa, Madrid
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario Clínico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Regional Universitario Carlos Haya, Málaga
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Virgen del Rocío, Seville
  - Hospital Universitario Dr. Peset, Valencia
  - Hospital Universitari i Politecnic La Fe, Valencia
  - Servicio de Neurología Hospital Viamed Montecanal., Zaragoza
- United Kingdom (7):
  - Ninewells Hospital, Dundee- Scotland, Dundee
  - Kings College Hospital, London
  - Charing Cross Hospital, London
  - Campus for Ageing and Vitality, Newcastle
  - Oxford University Hospitals NHS Foundation Trust, Oxford
  - North West Anglia NHS Foundation Trust, Peterborough
  - Derriford Hospital, Plymouth

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 586 participants with early-stage Parkinson's disease (PD) took part in the study across 110 investigative sites in 9 countries. The study consisted of double-blind treatment (DBT), where participants were randomized in 1:1 ratio to receive prasinezumab or placebo and an optional open-label extension (OLE).
Pre-assignment Details: After completing the DBT period, consenting & eligible participants entered the OLE period to receive prasinezumab. 3 participants in the prasinezumab arm and 1 participant in the placebo arm were randomized but not treated and 2 participants randomized to placebo arm received 1 dose of prasinezumab and were included in the prasinezumab arm for safety analysis. The study is still ongoing.
Groups:
- DBT Period: Placebo: Participants received prasinezumab matching placebo as an intravenous (IV) infusion, every 4 weeks (Q4W) up to at least 76 weeks.
- DBT Period: Prasinezumab: Participants received prasinezumab, 1500 milligrams (mg), as an intravenous (IV) infusion, Q4W up to at least 76 weeks.
- OLE Period: Prasinezumab: Eligible and consenting participants who completed the DBT period enrolled in the OLE period, to receive prasinezumab, 1500 mg, as an IV infusion, Q4W up to 104 weeks.
Period: DBT Period
Arm/Group | DBT Period: Placebo | DBT Period: Prasinezumab | OLE Period: Prasinezumab
Started | 293 | 293 | 0
Safety Analysis Set (SAS) (SAS included all participants who received at least one dose of study drug, with participants grouped according to treatment received.) | 290 (3 participants in prasinezumab arm and 1 participant in placebo arm were randomized but not treated. 2 participants randomized to placebo arm received 1 dose of prasinezumab and were included in the prasinezumab arm for safety analysis.) | 292 (3 participants in prasinezumab arm and 1 participant in placebo arm were randomized but not treated. 2 participants randomized to placebo arm received 1 dose of prasinezumab and were included in the prasinezumab arm for safety analysis.) | 0
Completed | 273 | 277 | 0
Not Completed | 20 | 16 | 0
Not completed — Death | 2 | 1 | 0
Not completed — Reason not Specified | 1 | 1 | 0
Not completed — Physician Decision | 4 | 0 | 0
Not completed — Withdrawal by Subject | 12 | 11 | 0
Not completed — Randomized but not Treated | 1 | 3 | 0
Period: OLE Period
Arm/Group | DBT Period: Placebo | DBT Period: Prasinezumab | OLE Period: Prasinezumab
Started | 0 | 0 | 534
Completed | 0 | 0 | 0
Not Completed | 0 | 0 | 534
Not completed — Ongoing in OLE | 0 | 0 | 534

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all randomized participants, with participants grouped according to their randomized treatment.
Groups:
- DBT Period: Placebo: Participants received prasinezumab matching placebo as an IV infusion, Q4W up to at least 76 weeks.
- DBT Period: Prasinezumab: Participants received prasinezumab, 1500 mg, as an IV infusion, Q4W up to at least 76 weeks.
- Total: Total of all reporting groups
Arm/Group | DBT Period: Placebo | DBT Period: Prasinezumab | Total
Number analyzed (Participants) | 293 | 293 | 586
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.4 (7.5) | 64.0 (7.2) | 64.2 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 104 | 110 | 214
  Male | 189 | 183 | 372
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 31 | 33 | 64
  Not Hispanic or Latino | 246 | 241 | 487
  Unknown or Not Reported | 16 | 19 | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 4 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 278 | 275 | 553
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 11 | 14 | 25

OUTCOME MEASURES:

1. Primary Outcome: DBT Period: Time to Confirmed Motor Progression Event Assessed by Movement Disorder Society - Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part III
Description: Time to confirmed motor progression event was the first time point of a worsening event defined as either >= 5 points increase in MDS-UPDRS Part III score (assessed in "OFF" medication state) from baseline sustained over 2 consecutive assessments or a change in medication after first occurrence of >= 5 points increase in MDS-UPDRS Part III score from baseline & before follow-up assessment. MDS-UPDRS Part III is a clinician rater scale that assessed the motor signs of PD. The scale is composed of 18 clinical domains or tasks, which yield 33 distinct scores or ratings. For each distinct rating, a numeric score is assigned between 0-4, where 0 = Normal, 1 = Slight, 2 = Mild, 3 = Moderate, and 4 = Severe. The total MDS-UPDRS Part III score (ranging from 0 to 132) is calculated by summing these 33 individual ratings, with higher scores indicating severe impairment.
Time Frame: From study start to end of DBT period to at least 76 weeks
Population: FAS included all randomized participants, with participants grouped according to their randomized treatment.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | DBT Period: Placebo | DBT Period: Prasinezumab
Number analyzed (Participants) | 293 | 293
weeks | 49.7 [40.1 to 58.1] | 61.1 [52.3 to 71.9]
Statistical Analysis 1: Comparison: DBT Period: Placebo vs DBT Period: Prasinezumab; Stratified Analysis; Test type: Superiority; p = 0.0657, Log Rank; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.69 to 1.01]

2. Secondary Outcome: DBT Period: Time-to-worsening of Participant's Motor Function as Reported by the Participant in the Presence of a Confirmed Motor Progression Event
Description: Time to worsening of the motor function was defined as ≥3 points increase in MDS-UPDRS Part II score from baseline in the presence of a confirmed motor progression event. For the confirmed motor progression event the definition is as per primary endpoint definition. MDS-UPDRS Part II assesses motor experiences of daily living & contained 13 questions answered by participant. For each question a numeric score is assigned between 0-4, 0 = Normal, 1=Slight, 2=Mild, 3=Moderate, 4=Severe. Score range: 0 to 52 with higher score=severe impairment.
Time Frame: From study start to end of DBT period to at least 76 weeks
Population: FAS included all randomized participants, with participants grouped according to their randomized treatment.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | DBT Period: Placebo | DBT Period: Prasinezumab
Number analyzed (Participants) | 293 | 293
weeks | 88.3 [62.7 to 105.1] | 112.1 [81.1 to NA] — Upper limit of 95 % confidence interval (CI) was not estimable due to insufficient follow-up duration to observe events and a very small number of individuals at risk by the end of the DBT period.
Statistical Analysis 1: Comparison: DBT Period: Placebo vs DBT Period: Prasinezumab; Test type: Superiority; p = 0.0914, Cox-regression adjusted; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.66 to 1.03]

3. Secondary Outcome: DBT Period: Time to Meaningful Worsening in Participant Global Impression of Change (PGI-C) Overall Disease Subscale
Description: The PGI is a measure commonly used in PD clinical trials to provide a concise assessment of overall health state. The change component (PGI-C) was intended to measure health state changes as reported by the participant on a 7-point scale (1=Very much improved to 7=Very much worse). The meaningfulness of the change was assessed and reported by the participant.
Time Frame: From study start to end of DBT period to at least 76 weeks
Population: FAS included all randomized participants, with participants grouped according to their randomized treatment.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | DBT Period: Placebo | DBT Period: Prasinezumab
Number analyzed (Participants) | 293 | 293
weeks | 36.1 [29.9 to 42.1] | 44.4 [38.1 to 52.1]
Statistical Analysis 1: Comparison: DBT Period: Placebo vs DBT Period: Prasinezumab; Test type: Superiority; p = 0.1574, Cox-regression adjusted; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.73 to 1.05]

4. Secondary Outcome: DBT Period: Time to Meaningful Worsening in Clinician Global Impression of Change (CGI-C) Overall Disease Subscale
Description: The CGI was a measure commonly used in PD clinical trials to provide a concise assessment of overall health state. The change component (CGI-C) was intended to measure health state changes as reported by the clinician on a 7-point scale (1=Very much improved to 7=Very much worse).
Time Frame: From study start to end of DBT period to at least 76 weeks
Population: FAS included all randomized participants, with participants grouped according to their randomized treatment.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | DBT Period: Placebo | DBT Period: Prasinezumab
Number analyzed (Participants) | 293 | 293
weeks | 52.1 [44.1 to 59.9] | 60.6 [56.1 to 67.3]
Statistical Analysis 1: Comparison: DBT Period: Placebo vs DBT Period: Prasinezumab; Test type: Superiority; p = 0.0622, Cox-regression adjusted; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.69 to 1.01]

5. Secondary Outcome: DBT Period: Time to Onset of Motor Complications as Assessed Through MDS-UPDRS Part IV
Description: MDS-UPDRS Part IV assessed motor complications of symptomatic treatment, dyskinesias, and motor fluctuations. The rater completed this assessment only for participants on L-Dopa treatment.
Time Frame: From study start to end of DBT period to at least 76 weeks
Population: FAS included all randomized participants, with participants grouped according to their randomized treatment.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | DBT Period: Placebo | DBT Period: Prasinezumab
Number analyzed (Participants) | 293 | 293
weeks | 91.1 [77.0 to 107.6] | 100.1 [81.0 to 117.1]
Statistical Analysis 1: Comparison: DBT Period: Placebo vs DBT Period: Prasinezumab; Test type: Superiority; p = 0.5515, Cox-regression adjusted; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.75 to 1.17]

6. Secondary Outcome: DBT Period: Change in Motor Function From Baseline to Week 76, as Measured by the MDS-UPDRS Part III Score
Description: MDS-UPDRS Part III is a clinician rater scale that assessed the motor signs of PD. The scale is composed of 18 clinical domains or tasks, which yield 33 distinct scores or ratings. For each distinct rating, a numeric score is assigned between 0-4, where 0 = Normal, 1 = Slight, 2 = Mild, 3 = Moderate, and 4 = Severe. The total MDS-UPDRS Part III score (ranging from 0 to 132) is calculated by summing these 33 individual ratings, with higher scores indicating severe impairment.
Time Frame: From baseline up to Week 76
Population: FAS included all randomized participants, with participants grouped according to their randomized treatment. Overall number analyzed is the number of participants with data available for analysis.
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | DBT Period: Placebo | DBT Period: Prasinezumab
Number analyzed (Participants) | 266 | 266
Units on a scale | 4.00 (0.592) | 3.61 (0.597)
Statistical Analysis 1: Comparison: DBT Period: Placebo vs DBT Period: Prasinezumab; Test type: Superiority; p = 0.5944, Mixed-model for Repeated Measures (MMRM); Difference in Adjusted Means = -0.39, 95% CI 2-sided [-1.84 to 1.05]

7. Secondary Outcome: DBT Period: Change in Bradykinesia and Rigidity From Baseline to Week 76, as Measured by the MDS-UPDRS Part III Bradykinesia and Rigidity Subscore
Description: MDS-UPDRS Part III is a clinician rater scale that assessed the motor signs of PD. The scale is composed of 18 clinical domains or tasks, which yield 33 distinct scores or ratings. For each distinct rating, a numeric score is assigned between 0-4, where 0 = Normal, 1 = Slight, 2 = Mild, 3 = Moderate, and 4 = Severe. For bradykinesia, subscore ranges from 0 to 52, while rigidity subscore ranges from 0 to 20, with higher scores indicating greater impairment. Change in bradykinesia and rigidity was assessed in "OFF" medication state. Adjusted mean is reported here.
Time Frame: From baseline up to Week 76
Population: as for outcome 6
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | DBT Period: Placebo | DBT Period: Prasinezumab
Number analyzed (Participants) | 267 | 266
Units on a scale | 2.77 (0.476) | 2.85 (0.479)
Statistical Analysis 1: Comparison: DBT Period: Placebo vs DBT Period: Prasinezumab; Test type: Superiority; p = 0.8955, MMRM; Difference in Adjusted Means = 0.08, 95% CI 2-sided [-1.08 to 1.24]

8. Secondary Outcome: DBT Period: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign (including abnormal laboratory values or abnormal clinical test results), symptoms, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. SAE is any significant hazard, contraindication, or side effect that is fatal or life-threatening, requires hospitalization or prolongation of an existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is medically significant or requires intervention. Number of participants with atleast 1 AE and SAE are reported here.
Time Frame: From study start to end of DBT period to at least 76 weeks
Population: Safety Analysis Set (SAS) included all participants who received at least one dose of study drug, with participants grouped according to treatment received. 3 participants in the prasinezumab arm and 1 participant in the placebo arm were randomized but not treated and 2 participants randomized to placebo arm received 1 dose of prasinezumab and were included in the prasinezumab arm for safety analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | DBT Period: Placebo | DBT Period: Prasinezumab
Number analyzed (Participants) | 290 | 292
Participants
  AEs | 260 | 267
  SAEs | 34 | 34

9. Secondary Outcome: DBT Period: Number of Participants With Adverse Events of Special Interest (AESI)
Description: An AE was any untoward medical occurrence in participant administered a pharmaceutical product & which does not necessarily have to have a causal relationship with treatment. It can therefore be any unfavorable and unintended sign (including abnormal laboratory values/ abnormal clinical test results), symptoms/disease temporally associated with use of pharmaceutical product, whether/not considered related to product. AESIs included potential drug-induced liver injury that include an elevated alanine transaminase (ALT) & aspartate aminotransferase (AST) in combination with either an elevated bilirubin/clinical jaundice defined by Hy's law and suspected transmission of an infectious agent by study drug.
Time Frame: From study start to end of DBT period to at least 76 weeks
Population: SAS included all participants who received at least one dose of study drug, with participants grouped according to treatment received. 3 participants in the prasinezumab arm and 1 participant in the placebo arm were randomized but not treated and 2 participants randomized to placebo arm received 1 dose of prasinezumab and were included in the prasinezumab arm for safety analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | DBT Period: Placebo | DBT Period: Prasinezumab
Number analyzed (Participants) | 290 | 292
Participants | 0 | 0

10. Secondary Outcome: DBT Period: Number of Participants With Treatment Discontinuation Due to AEs
Description: An AE was any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign (including abnormal laboratory values or abnormal clinical test results), symptoms, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product.
Time Frame: From study start to end of DBT period to at least 76 weeks
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | DBT Period: Placebo | DBT Period: Prasinezumab
Number analyzed (Participants) | 290 | 292
Participants | 3 | 2

11. Secondary Outcome: DBT Period: Number of Participants With Infusion Related Reactions (IRRs)
Description: IRRs were defined as any signs and symptoms (AEs) occurring during infusion and/or within 24 hours administration after the end of infusion and were considered related to study treatment by the investigator. Symptoms include flushing, rash, respiratory difficulty, hypotension, tachycardia.
Time Frame: From study start to end of DBT period to at least 76 weeks
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | DBT Period: Placebo | DBT Period: Prasinezumab
Number analyzed (Participants) | 290 | 292
Participants | 37 | 32

12. Secondary Outcome: DBT Period: Number of Participants With in Suicidal Ideation, as Measured by the Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: C-SSRS=assessment tool used to assess lifetime suicidality of participant (at baseline) as well as any new instances of suicidality (C-SSRS since last visit). Structured interview prompts recollection of suicidal ideation, including intensity of ideation, behavior, and attempts with actual/potential lethality. Categories have binary responses (yes/no) and include Wish to be Dead; Non-specific Active Suicidal Thoughts; Active Suicidal Ideation with Any Methods (Not Plan) without Intent to Act; Active Suicidal Ideation with Some Intent to Act, without Specific Plan; Active Suicidal Ideation with Specific Plan and Intent, Preparatory Acts and Behavior; Aborted Attempt; Interrupted Attempt; Actual Attempt (non-fatal); Completed Suicide. Suicidal ideation/behavior is indicated by a "yes" answer to any of the listed categories. Score of 0 is assigned if no suicide risk is present. Score of 1 or higher= suicidal ideation or behavior. Categories with non-zero values are only reported here.
Time Frame: From study start to end of DBT period to at least 76 weeks
Population: SAS included all participants who received at least one dose of study drug, with participants grouped according to treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | DBT Period: Placebo | DBT Period: Prasinezumab
Number analyzed (Participants) | 290 | 292
Participants
  Passive: Wish to be Dead | 6 | 5
  Non-specific Active Suicidal Thoughts | 2 | 2
  Active Suicidal Ideation with Any Methods (Not Plan) without Intent to Act | 3 | 0
  Self-injurious Behavior, no Suicidal Intent | 0 | 1

13. Secondary Outcome: DBT Period: Maximum Observed Concentration at Steady-state (Cmax,SS)
Time Frame: Day 1 of Weeks 1, 2, 4, 8, 12, 24, 36, 52, 64, 76
Population: Pharmacokinetic (PK) Analysis Set (PAS) included all randomized participants exposed to study treatment with sufficient dosing information and at least one adequately documented and quantifiable prasinezumab concentration.
Measure: Median (90% Confidence Interval); unit: micrograms/milliliter (µg/mL)
Arm/Group | DBT Period: Prasinezumab
Number analyzed (Participants) | 290
micrograms/milliliter (µg/mL) | 313.5 [217.3 to 514.9]

14. Secondary Outcome: DBT Period: Minimum Observed Concentration at Steady-state (Cmin,SS)
Time Frame: Day 1 of Weeks 1, 2, 4, 8, 12, 24, 36, 52, 64, 76
Population: PAS included all randomized participants exposed to study treatment with sufficient dosing information and at least one adequately documented and quantifiable prasinezumab concentration.
Measure: Median (90% Confidence Interval); unit: µg/mL
Arm/Group | DBT Period: Prasinezumab
Number analyzed (Participants) | 290
µg/mL | 28.7 [12.1 to 60.9]

15. Secondary Outcome: DBT Period: Area Under the Serum Concentration Time Curve Over the Dosing Interval (AUCTau,SS)
Time Frame: Day 1 of Weeks 1, 2, 4, 8, 12, 24, 36, 52, 64, 76
Population: as for outcome 14
Measure: Median (90% Confidence Interval); unit: hours*microgram/milliter (h*µg/mL)
Arm/Group | DBT Period: Prasinezumab
Number analyzed (Participants) | 290
hours*microgram/milliter (h*µg/mL) | 49384 [34850 to 82330]

16. Secondary Outcome: DBT Period: Percentage of Participants With Anti-Drug Antibodies (ADAs) at Baseline and Post-Treatment
Time Frame: From study start to end of DBT period to at least 76 weeks
Population: Immunogenicity population included all participants on active treatment with at least one ADA assessment. Percentages have been rounded off.
Measure: Number; unit: percentage of participants
Arm/Group | DBT Period: Prasinezumab
Number analyzed (Participants) | 289
percentage of participants | 0.3

17. Secondary Outcome: OLE Period: Number of Participants With AEs and SAEs
Description: An AE was any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign (including abnormal laboratory values or abnormal clinical test results), symptoms, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. SAE is any significant hazard, contraindication, or side effect that is fatal or life-threatening, requires hospitalization or prolongation of an existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is medically significant or requires intervention.
Time Frame: From signing of informed consent form up to 70 days after final dose of study treatment (Up to 66.6 months)
Reporting Status: Not Posted, anticipated posting 2027-12

18. Secondary Outcome: OLE Period: Number of Participants With AESI
Description: An AE was any untoward medical occurrence in participant administered a pharmaceutical product & which does not necessarily have to have a causal relationship with treatment. It can therefore be any unfavorable and unintended sign (including abnormal laboratory values/ abnormal clinical test results), symptoms/disease temporally associated with use of pharmaceutical product, whether/not considered related to product. AESIs included potential drug-induced liver injury that include an elevated ALT & AST in combination with either an elevated bilirubin/clinical jaundice defined by Hy's law and suspected transmission of an infectious agent by study drug.
Time Frame: From signing of informed consent form up to 70 days after final dose of study treatment (Up to 66.6 months)
Reporting Status: Not Posted, anticipated posting 2027-12

19. Secondary Outcome: OLE Period: Number of Participants With IRRs
Description: as for outcome 11
Time Frame: From signing of informed consent form up to 70 days after final dose of study treatment (Up to 66.6 months)
Reporting Status: Not Posted, anticipated posting 2027-12

20. Secondary Outcome: OLE Period: Number of Participants With in Suicidal Ideation, as Measured by the C-SSRS
Description: C-SSRS=assessment tool used to assess lifetime suicidality of participant (at baseline) as well as any new instances of suicidality (C-SSRS since last visit). Structured interview prompts recollection of suicidal ideation, including intensity of ideation, behavior, and attempts with actual/potential lethality. Categories have binary responses (yes/no) and include Wish to be Dead; Non-specific Active Suicidal Thoughts; Active Suicidal Ideation with Any Methods (Not Plan) without Intent to Act; Active Suicidal Ideation with Some Intent to Act, without Specific Plan; Active Suicidal Ideation with Specific Plan and Intent, Preparatory Acts and Behavior; Aborted Attempt; Interrupted Attempt; Actual Attempt (non-fatal); Completed Suicide. Suicidal ideation/behavior is indicated by a "yes" answer to any of the listed categories. Score of 0 is assigned if no suicide risk is present. Score of 1 or higher= suicidal ideation or behavior.
Time Frame: From signing of informed consent form up to 70 days after final dose of study treatment (Up to 66.6 months)
Reporting Status: Not Posted, anticipated posting 2027-12

ADVERSE EVENTS:
Time Frame: From study start until the end of DBT period for at least 76 weeks
Description: SAS included all participants who received at least one dose of study drug, with participants grouped according to treatment received. Data collected up to primary completion date is reported. Final data would be reported 1 year after study completion. 3 participants in the prasinezumab arm and 1 participant in the placebo arm were randomized but not treated and 2 participants randomized to placebo arm received 1 dose of prasinezumab and were included in the prasinezumab arm for safety analysis.
Arm/Group | DBT Period: Placebo | DBT Period: Prasinezumab
All-Cause Mortality (participants affected / at risk) | 2/290 | 1/292
Serious Adverse Events (participants affected / at risk) | 34/290 | 34/292
Other Adverse Events (participants affected / at risk) | 205/290 | 206/292
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DBT Period: Placebo (N=290) | DBT Period: Prasinezumab (N=292)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 4 (4)
Angina pectoris (Cardiac disorders) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Epiretinal membrane (Eye disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 3 (3) | 2 (2)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal food impaction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 1 (1)
Cyst (General disorders) | 1 (1) | 0 (0)
Infusion site reaction (General disorders) | 1 (1) | 0 (0)
Oedema (General disorders) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Endocarditis (Infections and infestations) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia influenzal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia pneumococcal (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 3 (3)
Urosepsis (Infections and infestations) | 1 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Shoulder fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebrospinal fluid leakage (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Migraine with aura (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Appendicectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DBT Period: Placebo (N=290) | DBT Period: Prasinezumab (N=292)
Constipation (Gastrointestinal disorders) | 15 (16) | 19 (26)
Diarrhoea (Gastrointestinal disorders) | 13 (17) | 15 (21)
Fatigue (General disorders) | 11 (11) | 21 (23)
COVID-19 (Infections and infestations) | 68 (77) | 84 (96)
Influenza (Infections and infestations) | 16 (16) | 21 (23)
Nasopharyngitis (Infections and infestations) | 31 (46) | 36 (48)
Upper respiratory tract infection (Infections and infestations) | 19 (21) | 21 (30)
Urinary tract infection (Infections and infestations) | 32 (44) | 24 (36)
Fall (Injury, poisoning and procedural complications) | 30 (60) | 34 (58)
Infusion related reaction (Injury, poisoning and procedural complications) | 36 (87) | 31 (55)
Arthralgia (Musculoskeletal and connective tissue disorders) | 25 (31) | 26 (37)
Back pain (Musculoskeletal and connective tissue disorders) | 40 (45) | 46 (66)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 18 (20) | 20 (22)
Dizziness (Nervous system disorders) | 18 (23) | 13 (17)
Headache (Nervous system disorders) | 18 (20) | 27 (45)
Anxiety (Psychiatric disorders) | 18 (18) | 17 (22)
Insomnia (Psychiatric disorders) | 16 (19) | 17 (19)
Hypertension (Vascular disorders) | 20 (21) | 14 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2025-04-15): https://cdn.clinicaltrials.gov/large-docs/31/NCT04777331/Prot_000.pdf
  • Statistical Analysis Plan (2024-08-05): https://cdn.clinicaltrials.gov/large-docs/31/NCT04777331/SAP_001.pdf